CLINICAL TRIAL: NCT06333730
Title: Comparison of Anesthetic Efficacy of Mental Nerve Block Versus Inferior Alveolar Nerve Block in Mandibular Anterior Teeth and Premolars in Symptomatic Irreversible Pulpitis- A Randomized Clinical Trial
Brief Title: Comparison of Anesthetic Efficacy of Mental Nerve Block Versus Inferior Alveolar Nerve Block in Mandibular Anterior Teeth and Premolars in Symptomatic Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prime Foundation (Other)
Responsible Party: Principal Investigator, Iftikhar Akbar, Head of Operative dentistry & Endodontic, Professor, Principal investigator, Prime Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PMC
Record Dates: First submitted 2023-10-31; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Symptomatic Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inferior Alveolar Nerve Block (IANB) (Experimental): 48 patients will be randomly selected in inferior alveolar nerve block group
  Interventions: Procedure: inferior alveolar nerve block
- Mental Nerve Block (MNB) (Experimental): 48 patients will be randomly selected in mental nerve block group
  Interventions: Procedure: mental nerve block

INTERVENTIONS:
Procedure: inferior alveolar nerve block — After informed consent, the needle will be inserted into the muco-buccal fold adjacent to the mandibular molars and advanced it towards the mandibular foramen, aiming slightly anteriorly and superiorly. Aspirating to check for blood or resistance, the needle will be repositioned if either was present. Once the needle will be correctly positioned, the dental practitioner will slowly inject 1.8-1.9 mL of the anesthetic solution.
  Arms: Inferior Alveolar Nerve Block (IANB)
Procedure: mental nerve block — After informed consent, the needle will be inserted into the buccal fold between the lower premolars. Aspirating to check for blood or resistance. Once needle is correctly positioned, 0.6-0.9 ml of the anesthetic solution will be deposited.
  Arms: Mental Nerve Block (MNB)

SUMMARY:
Symptomatic irreversible pulpitis is a painful condition that requires anesthesia to perform effective dental procedures. The mental nerve block and inferior alveolar nerve block are two commonly used techniques for achieving anesthesia in the mandibular teeth.

Study design: This randomized clinical trial study Number of participants: 96 participants which will be randomly divided into two groups: MINB and IANB.

Inclusion criteria: Participants with mandibular premolars or lower anterior experiencing sharp and persistent pain in response to thermal stimuli and an electric pulp tester, as well as bleeding during access opening, will be included.

Exclusion criteria: Participants with a medical history, allergies or contraindications to the local anesthetic, pregnant or breastfeeding women, those taking pain-affecting medication, or those experiencing pain in more than one tooth will be excluded.

Both techniques will use 2% lidocaine and adrenaline 1:80,000. Age, gender, and the efficacy of anesthesia will be recorded in both groups. The chi-square test will be used for comparison.

DETAILED DESCRIPTION:
Symptomatic irreversible pulpitis is a dental condition characterized by inflammation of the dental pulp, a soft tissue containing nerves and blood vessels located within the tooth's central cavity. The inflammation is severe and incapacitates the pulp's ability to heal naturally, leading to its eventual necrosis, hence the label "irreversible." The clinical manifestation of symptomatic irreversible pulpitis is excruciating, unrelenting pain, aggravated by exposure to hot or cold stimuli, and pressure. Inadequate intervention exposes the patient to the risk of infection or abscess formation, necessitating extensive dental procedures, including root canal therapy or tooth extraction.

The inferior alveolar nerve block (IANB) is a widely employed regional anesthesia technique in dentistry, utilized to provide profound anesthesia of the mandibular teeth and gingivae. It is a safe and reliable anesthesia technique commonly used in dentistry to prevent pain during procedures such as extractions, root canals, and implant placement, ensuring a comfortable experience for the patient. The mental or incisive nerve block is a dental anesthesia technique that anesthetizes the lower teeth, gums, lower lip, and chin by blocking the incisive and mental nerves, which are branches of the inferior alveolar nerve.

Local anesthesia in endodontics provides pain relief and patient comfort during procedures such as root canal therapy by blocking nerve impulses that transmit pain signals to the brain. Painful pulpitis may require pulpectomy under local anesthesia, but the effectiveness of injections can vary between teeth, with mandibular teeth being less responsive compared to maxillary teeth due to their thicker cortical bone and more complex anatomy. The inferior alveolar nerve is typically blocked in the lower molar and premolar region to achieve numbness. However, this approach may not always provide complete numbing of the nerve endings in the teeth. To enhance the likelihood of success, it is recommended to administer supplemental injections such as intra-osseous injections or applying 4% articaine through the cheek along with the inferior alveolar nerve block.

In a randomized clinical trial with 153 participants, the anesthetic success rates for mental nerve block and IANB were 53% and 47%, respectively, with no significant difference between them. However, combining both techniques by adding an IANB to MINB significantly improved the success rates to 82%. In a study conducted by Batista da Silva and colleagues, the effectiveness of 0.6 mL of 2% lidocaine and 4% articaine administered outside the mental foramen was evaluated. The results showed that using 4% articaine resulted in a 70% to 80% success rate for anesthesia.

This randomized clinical trial will be conducted at department of operative dentistry, Peshawar dental college, Peshawar. Ethical approval will be obtained from the hospital's ethical board. The sample size will be 96(48 in each group) at 5% level of significance, 80% power of test, using success for IANB to be 53% and to be mental block 80%. To participate in this study, patients needed to have exposed caries in their mandibular premolars or lower anterior causing sharp and persistent pain in response to thermal stimuli and an electric pulp tester, as well as bleeding during access opening. They also needed to have a medical history falling under American Society of Anesthesiologists class I or II and understand pain scales. Patients with allergies or contraindications to the local anesthetic, pregnant or breastfeeding women, those with a history of drug abuse, taking pain-affecting medication, or experiencing active pain in more than one tooth will be excluded.

The participants will be randomly divided into two, one receiving mental nerve block (MINB) and other IANB using block randomization technique. Each block size was eight. After obtaining informed consent, eligible patients will be randomly assigned to receive either mental nerve block or inferior alveolar nerve block. To perform an inferior alveolar block with 2% lidocaine and adrenaline 1:80,000, the dental practitioner will first explain the procedure to the patient and obtained their informed consent. The patient will be positioned comfortably in a dental chair and with their head supported. The injection site will be sterilized with an antiseptic solution, and the syringe will be loaded with the anesthetic solution. Next, the dental practitioner will inserted the needle into the mucobuccal fold adjacent to the mandibular molars and advanced it towards the mandibular foramen, aiming slightly anteriorly and superiorly. Aspirating to check for blood or resistance, the needle will be repositioned if either was present. Once the needle is correctly positioned, the dental practitioner slowly inject 1.8-1.9 mL of the anesthetic solution while checking for any signs of nerve stimulation, such as lip or tongue numbness. After completing the injection, the needle will be withdrawn and disposed of properly in a sharps container. For the mental block with 2% lidocaine and adrenaline 1:80,000, the mental foramen will be located, and the needle is inserted. After aspiration, 0.6-0.9 mL of anesthetic was injected while monitoring for nerve stimulation. The needle will then withdrawn and disposed of properly. After three minutes the anesthetic efficacy of each technique will be evaluated by assessing the pain score during access opening and instrumentation using a visual analog scale (10 point scale). Score more than 3 was considered ineffective.

The data analysis will be performed using SPSS version 22. Descriptive statistics will be calculated for all numeric and categorical data. The efficacy of two interventions (IANB and MINB) will be compared using the chi-square test. Stratification will be performed based on gender to control confounders. A significance level of P < 0.05 will be considered significance.

ELIGIBILITY:
Inclusion Criteria:

* Participants with mandibular premolars or lower anterior
* Experiencing sharp and persistent pain in response to thermal stimuli and an electric pulp tester
* Bleeding during access opening

Exclusion Criteria:

* Participants with a medical history
* Allergies or contraindications to the local anesthetic
* Pregnant or breastfeeding women
* Patient taking pain-affecting medication
* Patient experiencing pain in more than one tooth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
COMPARISON OF ANESTHETIC EFFICACY OF MENTAL NERVE BLOCK VERSUS INFERIOR ALVEOLAR NERVE BLOCK IN MANDIBULAR ANTERIORS TEETH AND PREMOLARS IN SYMPTOMATIC IRREVERSIBLE PULPITIS | Two months
  Pain after anesthesia in both groups will be assessed through Visual Pain analogue scale and greater than 3 will be considered ineffective

CONTACTS AND LOCATIONS:
Overall Officials: Saifa Rashad, BDS, Study Chair — Peshawar Dental College
Locations (1):
- Peshawar Dental College, Peshawar, Khyber Pakhtunkhwa, Pakistan